CLINICAL TRIAL: NCT00688792
Title: Reasons for Poor Adherence for Long-Term Preventing Therapy in Children With Asthma
Brief Title: Maternal Variables Associated With Adherence in Children With Asthma
Acronym: asthma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Prof. Dan Engelhard, MD, Hadassah Medical Organization
Other Study IDs: asthma1-HMO-CTIL
Record Dates: First submitted 2008-05-29; First posted 2008-06-03 (Estimated); Last update posted 2008-06-03 (Estimated); Status verified 2008-05

CONDITIONS: Asthma
Keywords: Asthma; Children; Adherence; Maternal factors
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
A questionnaire will be used in order to find out the reasons for poor adherence for long-term treatment in children with asthma. The hypotheses is maternal factors including the knowledge that asthma is a chronic disease and fear to administer inhaled steroids are major obstacles for appropriate adherence.

DETAILED DESCRIPTION:
Parents to children aged 2 - 12 years with moderate to severe asthma who need long-term treatment with inhaled steroids will be included in the study. Three weeks after their visit in the clinic, they will be requested to answer a questionnaire by telephone.

ELIGIBILITY:
Inclusion Criteria:

* Parents to children aged 2 - 12 years with moderate to severe asthma to whom inhaled steroids was described for a period of at least 4 weeks.

Exclusion Criteria:

* Parents who will not agree to sign the consent form and parents who do not speak and understand the Hebrew language.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Parents to children aged 2 - 12 years with moderate to severe asthma.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2008-07; Primary Completion 2010-06 (Estimated); Study Completion 2011-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Dan Engelhard, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel